CLINICAL TRIAL: NCT05093205
Title: A PHASE 1, OPEN-LABEL, TWO-PART STUDY TO EVALUATE THE EFFECT OF TWO STEADY-STATE DOSE LEVELS OF PF-06882961 ON THE PHARMACOKINETICS OF SINGLE ORAL DOSES OF ATORVASTATIN AND MIDAZOLAM IN HEALTHY ADULTS AND AN ORAL CONTRACEPTIVE IN HEALTHY POST-MENOPAUSAL FEMALES
Brief Title: STUDY TO EVALUATE THE EFFECT OF PF-06882961 ON SINGLE DOSE ATORVASTATIN, MEDAZOLAM AND ORALCONTRACEPTIVE PHARMACOKINETICS IN HEALTHY ADULT PARTICIPANTS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: C3421047
Record Dates: First submitted 2021-10-13; First posted 2021-10-26 (Actual); Results first posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-03

CONDITIONS: Healthy Adults
MeSH Terms: interventions — danuglipron; Atorvastatin; Midazolam; Ethinyl Estradiol-Norgestrel Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental): To evaluate the effect of 2 steady-state dose levels of PF-06882961 on the Single Dose pharmacokinetics of atorvastatin (20 mg tablet) and midazolam (5 mg syrup).
  Interventions: Drug: PF-06882961; Drug: Atorvastatin; Drug: Midazolam
- Part B (Experimental): To evaluate the effect of 2 steady-state dose levels of PF-06882961 on the Single Dose pharmacokinetics of an Oral Contraceptive (Levonorgestrel 0.15 mg and Ethinyl Estradiol 0.03 mg tablet).
  Interventions: Drug: PF-06882961; Drug: Levonorgestrel & Ethinyl Estradiol

INTERVENTIONS:
Drug: PF-06882961 — Tablets
Drug: Atorvastatin — Tablets
  Arms: Part A
Drug: Midazolam — Syrup
  Arms: Part A
Drug: Levonorgestrel & Ethinyl Estradiol — Tablet
  Arms: Part B

SUMMARY:
The purpose of this study is to characterize the effect of PF-06882961, administered at 2 steady-state dose levels, on the PK of single doses of atorvastatin (20 mg) or midazolam (5 mg), administered separately, in healthy adult male and female participants (Part A), or an OC in healthy PM female participants (Part B).

ELIGIBILITY:
Inclusion Criteria:

* Part A Only - Healthy male and female participants must be 18 to 65 years of age, inclusive, at the time of signing the ICD (healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, physical examination, including blood pressure and pulse rate measurement, standard 12 lead ECG and clinical laboratory tests).
* Part B Only - Healthy PM female participants between 40 and 65 years of age, inclusive, at the time of signing the ICD (healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, physical examination, including BP and PR measurement, standard 12 lead ECG and clinical laboratory tests). Subjects must be amenorrheic for at least 12 months. Women who are 60 years of age or younger must also have an FSH that is within the laboratory's reference range for PM women.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* BMI- 20.0 kg/m2 to <30.0 kg/m2 at Screening.
* Stable body weight, defined as <5 % change (per participant report) for 90 days before Screening.
* Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, prior bariatric surgery, gastrectomy, or any area of intestinal resection, active inflammatory bowel disease or pancreatic insufficiency).
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Known intolerance or hypersensitivity to GLP-1R agonists.
* Known hypersensitivity to atorvastatin or midazolam (for participants in Part A), or LE and EE (for participants in Part B).
* Personal or family history of MTC or MEN2 or study participants with suspected MTC per the investigator's judgment.
* Symptomatic gallbladder disease.
* History of major depressive disorder or history of other severe psychiatric disorders (eg, schizophrenia or bipolar disorder) within the last 2 years from screening.
* Any lifetime history of a suicide attempt.
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study intervention.
* Systemic therapy with any of the medications that are moderate or strong CYP3A4/5, CYP2C9 and/or CYP2C19 inhibitors within 28 days or 5 half-lives (whichever is longer) or moderate or strong CYP3A, CYP2C9 and/or CYP2C19 inducers within 28 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention.
* Systemic therapy with inhibitors of the BCRP transporter within 28 days or 5 half lives (whichever is longer) prior to the first dose of study intervention.
* Current use of any prohibited concomitant medication(s) or those unwilling/unable to use a permitted concomitant medication(s).
* Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of study intervention used in this study (whichever is longer).
* Known prior participation in a trial involving PF-06882961.
* A PHQ-9 score ≥15 obtained at Screening or Day -1 in Study.
* Response of "yes" to question 4 or 5, or on any suicidal behavioral question on the C SSRS at Screening or Day -1 in Study.
* A positive urine drug test.
* Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest. BP should be measured in triplicate and the average of the 3 BP values should be used to determine the participant's eligibility. Note: At screening, the participant's arm circumference should be measured (eg, using a flexible anthropometric tape) at the midpoint of the length of the upper arm and the appropriate cuff selected and used throughout the study.
* Screening 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, QTcF interval >450 msec, complete LBBB, signs of an acute or indeterminate age myocardial infarction, ST-T interval changes suggestive of myocardial ischemia, second or third degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If QTcF exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTcF or QRS values should be used to determine the participant's eligibility. Computer interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding participants.
* Participants with ANY of the following abnormalities in clinical laboratory tests at Screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

  * HbA1c ≥6.5%.
  * Aspartate AST or ALT level ≥2 times the ULN.
  * Total bilirubin level ≥1.5 times the ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN.
  * TSH >1.5x the ULN or <LLN.
  * Serum calcitonin > the ULN.
  * Amylase or lipase > the ULN.
  * Fasting blood glucose ≥126 mg/dL.
  * Fasting C-peptide <0.8 ng/mL.
  * eGFR <70 mL/min/1.73 m2 as calculated by the CKD-EPI equation.
  * Positive testing for HIV, HepBsAg, or HCVAb. Study participants positive for HCVAb are to be excluded unless known to have been treated with a known curative therapy and negative for HCV RNA. Hepatitis B vaccination is allowed.
  * A positive SARS-CoV-2 test.
* Participation in a formal weight reduction program (eg, Weight Watchers) within 90 days prior to Screening.
* History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit or 3 ounces (90 mL) of wine).
* Current use of tobacco or nicotine containing products in excess of the equivalent of 5 cigarettes per day.
* Known or suspected illicit drug use.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing randomization (Day-1).
* History of sensitivity to heparin or heparin induced thrombocytopenia if Hep-lock is used for IV blood draw.
* Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
* Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2022-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Anaheim Clinical Trials, LLC, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3421047

RESULTS

PARTICIPANT FLOW:
Groups:
- Atorvastatin 20 mg (Part A Period 1): Participants received single dose of atorvastatin 20 mg orally on Day 1 in Part A Period 1.
- Midazolam 5 mg (Part A Period 2): Participants received single dose of midazolam 5 mg orally on Day 1 of Period 2 in Part A.
- PF-06882961 Titration up to 120 mg BID (Part A Period 3): Participants received PF-06882961 10 mg BID on Days 1-4, 20 mg BID on Days 5-8, 40 mg BID on Days 9-12, 60 mg BID on Days 13-16, 80 mg BID on Days 17-20, 100 mg BID on Days 21-24, and 120 mg BID on Days 25-31 of Period 3.
- PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4): Participants received PF-06882961 120 mg BID + atorvastatin 20 mg SD on Day 1 of Period 4 and PF-06882961 120 mg BID on Days 2-3 of Period 4.
- PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5): Participants received PF-06882961 120 mg BID + midazolam 5 mg SD on Day 1 of Period 5 in Part A.
- PF-06882961 Titration up to 200 mg BID (Part A Period 6): Participants received PF-06882961 140 mg BID on Days 1-4, 160 mg BID on Days 5-8, 180 mg BID on Days 9-12, and 200 mg BID on Days 13-19 of Period 6 in Part A.
- PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7): Participants received PF-06882961 200 mg BID + atorvastatin 20 mg SD on Day 1 of Period 7 and PF-06882961 200 mg BID on Days 2-3 of Period 7 in Part A.
- PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8): Participants received PF-06882961 200 mg BID + midazolam 5 mg SD on Day 1 of Period 8 in Part A.
- 0.15 mg LE & 0.03 mg EE (Part B Period 1): Participants received single dose of oral contraceptive on Day 1 of Period 1 in Part B.
- PF-06882961 Titration up to 120 mg BID (Part B Period 2): Participants received PF-06882961 10 mg BID on Days 1-4, 20 mg BID on Days 5-8, 40 mg BID on Days 9-12, 60 mg BID on Days 13-16, 80 mg BID on Days 17-20, 100 mg BID on Days 21-24, and 120 mg BID on Days 25-31 of Period 2 in Part B.
- PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3): Participants received PF-06882961 120 mg BID + OC SD on Day 1 and PF-06882961 120 mg BID on Days 2-5 of Period 3 in Part B.
- PF-06882961 Titration up to 200 mg BID (Part B Period 4): Participants received PF-06882961 140 mg BID on Days 1-4, 160 mg BID on Days 5-8, 180 mg BID on Days 9-12, and 200 mg BID on Days 13-19 of Period 4 in Part B.
- PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5): Participants received PF-06882961 200 mg BID + oral contraceptive SD on Day 1 and PF-06882961 200 mg BID on Days 2-5 of Period 5 in Part B.
Period: Part A Period 1 - Treatment
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8) | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Started | 18 | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".)
Completed | 18 | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Period 1 - Follow-Up
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8) | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Started | 15 | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".)
Completed | 15 | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".) | 0 (This period only applies to the group "Part A Period 1".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Period 2 - Treatment
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8) | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Started | 0 (This period only applies to the group "Part A Period 2".) | 18 | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".)
Completed | 0 (This period only applies to the group "Part A Period 2".) | 17 | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".)
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Period 2 - Follow-Up
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8) | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Started | 0 (This period only applies to the group "Part A Period 2".) | 15 | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".)
Completed | 0 (This period only applies to the group "Part A Period 2".) | 15 | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".) | 0 (This period only applies to the group "Part A Period 2".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Period 3 - Treatment
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8) | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Started | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 17 | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".)
Completed | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 13 | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".)
Not Completed | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Period 3 - Follow-Up
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8) | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Started | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 15 | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".)
Completed | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 15 | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".) | 0 (This period only applies to the group "Part A Period 3".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Period 4 - Treatment
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8) | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Started | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 13 | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".)
Completed | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 13 | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Period 4 - Follow-Up
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8) | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Started | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 13 | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".)
Completed | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 13 | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".) | 0 (This period only applies to the group "Part A Period 4".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Period 5 - Treatment
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8) | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Started | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 13 | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".)
Completed | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 13 | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Period 5 - Follow-Up
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8) | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Started | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 13 | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".)
Completed | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 13 | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".) | 0 (This period only applies to the group "Part A Period 5".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Period 6 - Treatment
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8) | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Started | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 13 | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".)
Completed | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 6 | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Period 6 - Follow-Up
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8) | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Started | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 13 | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".)
Completed | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 13 | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".) | 0 (This period only applies to the group "Part A Period 6".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Period 7 - Treatment
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8) | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Started | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 5 | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".)
Completed | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 5 | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Period 7 - Follow-Up
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8) | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Started | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 5 | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".)
Completed | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 5 | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".) | 0 (This period only applies to the group "Part A Period 7".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Period 8 - Treatment
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8) | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Started | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 6 | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".)
Completed | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 5 | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Part A Period 8 - Follow-Up
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8) | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Started | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 6 | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".)
Completed | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 6 | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".) | 0 (This period only applies to the group "Part A Period 8".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B Period 1 - Treatment
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8) | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Started | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 17 | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".)
Completed | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 16 | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Part B Period 1 - Follow-Up
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8) | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Started | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 15 | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".)
Completed | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 15 | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".) | 0 (This period only applies to the group "Part B Period 1".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B Period 2 - Treatment
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8) | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Started | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 16 | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".)
Completed | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 14 | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Period: Part B Period 2 - Follow-Up
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8) | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Started | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 15 | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".)
Completed | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 14 | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".) | 0 (This period only applies to the group "Part B Period 2".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Part B Period 3 - Treatment
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8) | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Started | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 14 | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".)
Completed | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 12 | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Period: Part B Period 3 - Follow-Up
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8) | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Started | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 13 | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".)
Completed | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".) | 11 | 0 (This period only applies to the group "Part B Period 3".) | 0 (This period only applies to the group "Part B Period 3".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Period: Part B Period 4 - Treatment
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8) | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Started | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 12 | 0 (This period only applies to the group "Part B Period 4".)
Completed | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 9 | 0 (This period only applies to the group "Part B Period 4".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Period: Part B Period 4 - Follow-Up
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8) | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Started | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 11 | 0 (This period only applies to the group "Part B Period 4".)
Completed | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 0 (This period only applies to the group "Part B Period 4".) | 10 | 0 (This period only applies to the group "Part B Period 4".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Part B Period 5 - Treatment
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8) | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Started | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 9
Completed | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B Period 5 - Follow-Up
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8) | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Started | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 9
Completed | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 0 (This period only applies to the group "Part B Period 5".) | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of study intervention
Groups:
- All Participants in Part A: Participants underwent Period 1 to 8 and received study interventions as follows: Period 1: atorvastatin 20mg single dose (SD) on Day 1; Period 2: midazolam 5mg SD on Day 1; Period 3: PF-06882961 10mg twice daily (BID) on Days 1-4, 20mg BID on Days 5-8, 40mg BID on Days 9-12, 60mg BID on Days 13-16, 80mg BID on Days 17-20, 100mg BID on Days 21-24, and 120mg BID on Days 25-31; Period 4: PF-06882961 120mg BID+atorvastatin SD on Day 1, PF-06882961 120mg on Days 2-3; Period 5: PF-06882961 120 mg BID+ midazolam SD on Day 1; Period 6: PF-06882961 140 mg BID on Days 1-4, 160 mg BID on Days 5-8, 180 mg BID on Days 9-12, 200 mg BID on Days 13-19; Period 7: PF-06882961 200 mg BID+atorvastatin SD on Day 1, PF-06882961 200 mg BID on Days 2-3; Part 8: PF-06882961 200 mg BID+ midazolam SD on Day 1.
- All Participants in Part B: Participants underwent Period 1 to 5 and received study interventions as follows: Period 1: oral contraceptive (OC) SD on Day 1; Period 2:PF-06882961 10mg BID on Days 1-4, 20mg BID on Days 5-8, 40mg BID on Days 9-12, 60mg BID on Days 13-16, 80mg BID on Days 17-20, 100mg BID on Days 21-24, and 120mg BID on Days 25-31; Period 3: PF-06882961 120mg BID+OC SD on Day 1, PF-06882961 120mg on Days 2-5; Period 4: PF-06882961 140 mg BID on Days 1-4, 160 mg BID on Days 5-8, 180 mg BID on Days 9-12, 200 mg BID on Days 13-19; Period 5: PF-06882961 200 mg BID+OC SD on Day 1, PF-06882961 200 mg BID on Days 2-5.
- Total: Total of all reporting groups
Arm/Group | All Participants in Part A | All Participants in Part B | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Mean (SD) | 41.2 (11.63) | 54.5 (4.16) | 47.7 (11.01)
Age, Customized [Number; unit: Participants]
  <18 Years | 0 | 0 | 0
  18-25 Years | 2 | 0 | 2
  26-35 Years | 4 | 0 | 4
  36-45 Years | 4 | 0 | 4
  >45 Years | 8 | 17 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 17 | 19
  Male | 16 | 0 | 16
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 15 | 14 | 29
  Black or African American | 2 | 2 | 4
  Asian | 1 | 1 | 2
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 8 | 9 | 17
  Not Hispanic or Latino | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: (Part A) Area Under the Concentration-time Curve From Time 0 to Infinity (AUCinf) of Atorvastatin in Periods 1, 4, and 7
Description: Atorvastatin was given on Day 1 in Periods 1, 4 and 7 of Part A and blood samples were collected for atorvastatin pharmacokinetic (PK) at the preset time points described in the Time Frame. AUCinf calculated area under the plasma concentration-time profile from time 0 extrapolated to infinite time.
Time Frame: For Part A Periods 1, 4, and 7: At 0 (prior to atorvastatin dose), 0.5, 1, 1.5, 2, 4, 6, 9, 12, 24, 36, 48, 72 hours (only Periods 1 & 4) post atorvastatin dose on Day 1 of each period.
Population: Only participants with evaluable results for the pharmacokinetic (PK) parameter were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7)
Number analyzed (Participants) | 16 | 11 | 3
nanogram*hour/milliliter (ng*hr/mL) | 32.27 (41) | 46.94 (72) | 54.43 (22)

2. Primary Outcome: (Part A) AUCinf of Midazolam in Periods 2, 5, and 8
Description: Midazolam was given on Day 1 in Periods 2, 5 and 8 of Part A and blood samples were collected for midazolam PK at the preset time points described in the Time Frame. AUCinf calculated area under the plasma concentration-time profile from time 0 extrapolated to infinite time.
Time Frame: For Part A Periods 2, 5, and 8: At 0 (prior to midazolam dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hours (only for Periods 2 & 5) post midazolam dose on Day 1 of each period.
Population: Only participants with evaluable results for the PK parameter were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Midazolam 5 mg (Part A Period 2) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8)
Number analyzed (Participants) | 18 | 13 | 5
ng*hr/mL | 70.53 (32) | 58.81 (40) | 49.78 (22)

3. Primary Outcome: (Part B) AUCinf of Levonorgestrel in Periods 1, 3 and 5
Description: Levonorgestrel was given on Day 1 in Periods 1, 3 and 5 of Part B and blood samples were collected for levonorgestrel PK at the preset time points described in the Time Frame. AUCinf calculated area under the plasma concentration-time profile from time 0 extrapolated to infinite time.
Time Frame: For Part B Periods 1, 3, 5: At 0 (prior to levonorgestrel dose), 0.5, 1, 1.5, 2, 4, 8, 12, 24, 48, 72, 96, 120 hours post levonorgestrel dose on Day 1 of each period.
Population: Only participants with evaluable results for the PK parameter were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram*hour/milliliter (pg*hr/mL)
Arm/Group | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Number analyzed (Participants) | 15 | 12 | 8
picogram*hour/milliliter (pg*hr/mL) | 48800 (42) | 62330 (61) | 66490 (57)
Statistical Analysis 1: Comparison: 0.15 mg LE & 0.03 mg EE (Part B Period 1) vs PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3); Test type: Other — 0.15 mg LE & 0.03 mg EE was the Reference treatment (Part B Period 1), PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE was the Test treatment (Period 3); Mixed Models Analysis; Specified in comments = 122.48, 90% CI 2-sided [106.96 to 140.25] — A mixed effects model with treatment as a fixed effect and participant as a random effect was used was applied to calculate the ratio (Test/Reference) of adjusted means and 90% CIs for Ratio. The ratio (and 90% CI) is expressed as percentage
Statistical Analysis 2: Comparison: 0.15 mg LE & 0.03 mg EE (Part B Period 1) vs PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5); Test type: Other — 0.15 mg LE & 0.03 mg EE was the Reference treatment (Part B Period 1), PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE was the Test treatment (Period 5); Mixed Models Analysis; Specified in comments = 143.83, 90% CI 2-sided [122.64 to 168.68] — [estimate comment as in outcome 3, analysis 1]

4. Primary Outcome: (Part B) AUCinf of Ethinyl Estradiol in Periods 1, 3 and 5
Description: Ethinyl estradiol (EE) was given on Day 1 in Periods 1, 3 and 5 of Part B and blood samples were collected for ethinyl estradiol PK at the preset time points described in the Time Frame. AUCinf calculated area under the plasma concentration-time profile from time 0 extrapolated to infinite time.
Time Frame: For Part B Periods 1, 3, 5: At 0 (prior to EE dose), 0.5, 1, 1.5, 2, 4, 8, 12, 24, 48, 72, 96, 120 hours post EE dose on Day 1 in Periods 1, 3, 5 of each period.
Population: Only participants with evaluable results for the PK parameter were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*hr/mL
Arm/Group | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Number analyzed (Participants) | 16 | 12 | 9
pg*hr/mL | 772.1 (41) | 723.5 (24) | 604.4 (33)
Statistical Analysis 1: Comparison: 0.15 mg LE & 0.03 mg EE (Part B Period 1) vs PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3); Test type: Other — [test comment as in outcome 3, analysis 1]; Mixed Models Analysis; Specified in comments = 104.46, 90% CI 2-sided [92.56 to 117.89] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: 0.15 mg LE & 0.03 mg EE (Part B Period 1) vs PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5); Test type: Other — [test comment as in outcome 3, analysis 2]; Mixed Models Analysis; Specified in comments = 92.77, 90% CI 2-sided [81.05 to 106.19] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: (Part A) Number of Participants With Treatment Emergent Adverse Events (TEAE) During Part A of the Study
Description: An AE was any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An serious adverse event was defined as any untoward medical occurrence that,at any dose:resulted in death;was life-threatening;required inpatient hospitalization or prolongation of existing hospitalization;resulted in persistent disability/incapacity; was a congenital anomaly/birth defect;or other serious situations such as important medical events. The investigator was required to use clinical judgment to assess the potential relationship between investigational product and each AE, to define an treatment-related AE.
Time Frame: From Baseline up to follow-up telephone contact (Days 90-97) in Part A of the study.
Population: All participants randomly assigned to study intervention and who had at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8)
Number analyzed (Participants) | 18 | 18 | 17 | 13 | 13 | 13 | 5 | 6
Participants
  Participants with adverse events | 2 | 3 | 13 | 5 | 4 | 12 | 5 | 2
  Participants with serious adverse events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participants with severe adverse events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participants discontinued from study due to AEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participants discontinued study drug due to AE and continue study | 0 | 0 | 2 | 0 | 0 | 7 | 0 | 1
  Participants with dose reduced or temporary discontinuation due to AE | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 0

6. Secondary Outcome: (Part B) Number of Participants With TEAE During Part B of the Study
Description: as for outcome 5
Time Frame: From Baseline up to follow-up telephone contact (Days 94-101) in Part B of the study.
Population: All participants randomly assigned to study intervention and who had at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Number analyzed (Participants) | 17 | 16 | 14 | 12 | 9
Participants
  Participants with adverse events | 5 | 15 | 7 | 12 | 7
  Participants with serious adverse events | 0 | 0 | 0 | 0 | 0
  Participants with severe adverse events | 0 | 0 | 0 | 0 | 0
  Participants discontinued from study due to AEs | 0 | 0 | 0 | 0 | 0
  Participants discontinued study drug due to AE and continue study | 0 | 2 | 2 | 2 | 0
  Participants with dose reduced or temporary discontinuation due to AE | 0 | 2 | 0 | 2 | 0

7. Secondary Outcome: (Part A) Number of Participants With Clinical Laboratory Abnormalities During Part A of the Study (Without Regard to Baseline Abnormality)
Description: Laboratory tests (including hematology, clinical chemistry, urinalysis) were reported and abnormalities were defined for laboratory values that met specific criteria.
Time Frame: From Baseline up to follow-up visit (Days 69-72) in Part A of the study.
Population: All participants randomly assigned to study intervention and who had at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Atorvastatin 20 mg (Part A Period 1): Participants received single dose of atorvastatin 20 mg orally on Day 1 of Period 1 in Part A.
- PF-06882961 Titration up to 120 mg BID (Part A Period 3): Participants received PF-06882961 10 mg BID on Days 1-4, 20 mg BID on Days 5-8, 40 mg BID on Days 9-12, 60 mg BID on Days 13-16, 80 mg BID on Days 17-20, 100 mg BID on Days 21-24, and 120 mg BID on Days 25-31 of Period 3 in Part A.
- PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4): Participants received PF-06882961 120 mg BID + atorvastatin 20 mg SD on Day 1 of Period 4 and PF-06882961 120 mg BID on Days 2-3 of Period 4 in Part A.
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8)
Number analyzed (Participants) | 18 | 18 | 17 | 13 | 13 | 13 | 5 | 6
Participants | 0 | 15 | 16 | 2 | 5 | 12 | 0 | 6

8. Secondary Outcome: (Part B) Number of Participants With Clinical Laboratory Abnormalities During Part B of the Study (Without Regard to Baseline Abnormality)
Description: as for outcome 7
Time Frame: From Baseline up to follow-up visit (Days 72-75) in Part B of the study.
Population: All participants randomly assigned to study intervention and who had at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- PF-06882961 Titration up to 120 mg BID (Period 2): Participants received PF-06882961 10 mg BID on Days 1-4, 20 mg BID on Days 5-8, 40 mg BID on Days 9-12, 60 mg BID on Days 13-16, 80 mg BID on Days 17-20, 100 mg BID on Days 21-24, and 120 mg BID on Days 25-31 of Period 2 in Part B.
Arm/Group | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Number analyzed (Participants) | 17 | 16 | 4 | 12 | 9
Participants | 17 | 16 | 2 | 12 | 9

9. Secondary Outcome: (Part A) Number of Participants With Vital Signs Abnormalities During Part A of the Study
Description: Supine blood pressure (mm Hg) and pulse rate (beats per minute) were measured. Supine BP was measured with the participant's arm supported at heart level and recorded to the nearest mmHg after approximately 5 minutes of rest.
Time Frame: From Baseline up to follow-up visit (Days 69-72) in Part A of the study.
Population: All participants randomly assigned to study intervention and who had at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8)
Number analyzed (Participants) | 18 | 18 | 17 | 13 | 13 | 13 | 5 | 6
Participants
  Supine systolic blood pressure (SBP) value <90 mm Hg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine SBP change >=30 mm Hg increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine SBP change >=30 mm Hg decrease | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 1
  Supine diastolic blood pressure (DBP) value <50 mm Hg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine DBP >= 20 mm Hg increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Supine DBP >= 20 mm Hg decrease | 1 | 1 | 2 | 2 | 3 | 1 | 2 | 1
  Pulse rate value <40 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse rate value >120 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: (Part B) Number of Participants With Vital Signs Abnormalities During Part B of the Study
Description: Supine blood pressure (mm Hg) and pulse rate (bpm) were measured. Supine BP was measured with the participant's arm supported at heart level and recorded to the nearest mmHg after approximately 5 minutes of rest.
Time Frame: From Baseline up to follow-up visit (Days 72-75) in Part B of the study.
Population: All participants randomly assigned to study intervention and who had at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Number analyzed (Participants) | 17 | 16 | 2 | 12 | 9
Participants
  Supine SBP value <90 mm Hg | 0 | 0 | 0 | 0 | 0
  Supine SBP change >=30 mm Hg increase | 0 | 0 | 0 | 0 | 0
  Supine SBP change >=30 mm Hg decrease | 1 | 1 | 0 | 1 | 1
  Supine DBP value <50 mm Hg | 0 | 0 | 0 | 0 | 0
  Supine DBP >= 20 mm Hg increase | 0 | 0 | 0 | 0 | 0
  Supine DBP >= 20 mm Hg decrease | 1 | 3 | 0 | 1 | 1
  Pulse rate value <40 bpm | 0 | 0 | 0 | 0 | 0
  Pulse rate value >120 bpm | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: (Part A) Percentage of Change From Baseline in Body Weight
Description: Percentage of changes from Baseline in body weight of the participants were measured.
Time Frame: Percentage of change from Baseline 1: from the last pre-dose measurement in Part A Period 1 (ie, Baseline 1) to Day 2 of Part A Period 8; percentage of Change from the last predose measurement in Part A Period 3 (ie, Baseline 2) to Day 2 of Period 8.
Population: All participants who were randomly assigned to study intervention and had at least 1 dose of study intervention, and with evaluable body weight measurement were included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | All Participants in Part A
Number analyzed (Participants) | 6
percentage
  Baseline 1 - Period 8 Day 2 / PF-06882961 200 mg BID + Midazolam 5 mg | -9.04 (3.539)
  Baseline 2 - Period 8 Day 2 / PF-06882961 200 mg BID + Midazolam 5 mg | -9.30 (4.159)

12. Secondary Outcome: (Part B) Percentage of Change From Baseline in Body Weight
Description: Percentage of changes from Baseline in body weight of the participants were measured.
Time Frame: Percentage of Change from Baseline 1:from the last pre-dose measurement in Part B Period 1 (ie, Baseline 1) to Day 2 of Part B Period 8;percentage of Change from the last predose measurement in Part B Period 2 (ie, Baseline 2) to Day 6 of Part B Period 5.
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | All Participants in Part B
Number analyzed (Participants) | 17
percentage
  Baseline 1 - Period 5 Day 6 / PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE: number analyzed (Participants) | 9
  Baseline 1 - Period 5 Day 6 / PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE | -8.77 (2.190)
  Baseline 2 - Period 5 Day 6 / PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE: number analyzed (Participants) | 9
  Baseline 2 - Period 5 Day 6 / PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE | -5.40 (1.503)

13. Secondary Outcome: (Part A) Number of Participants With Treatment Emergent Electrocardiograms (ECG) Abnormalities During Part A of the Study
Description: Standard 12-lead ECGs utilizing limb leads were collected using an ECG machine that automatically calculated the heart rate and measured PR, QT, and QT interval corrected for heart rate (QTc) and QRS complex.
Time Frame: From Baseline up to follow-up visit (Days 69-72) in Part A of the study.
Population: All participants randomly assigned to study intervention and who had at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8)
Number analyzed (Participants) | 18 | 18 | 17 | 13 | 13 | 13 | 5 | 6
Participants
  PR interval value >=300 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR interval %change >=25/50% msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QRS interval value >= 140 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QRS interval %change >=50% msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF 450 msec < value <=480 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF 480 msec < value <=500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF value >500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF 30 msec < change <=60 msec | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 1
  QTcF change >60 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: (Part B) Number of Participants With Treatment Emergent ECG Abnormalities During Part B of the Study
Description: as for outcome 13
Time Frame: From Baseline up to follow-up visit (Days 72-75) in Part B of the study.
Population: All participants randomly assigned to study intervention and who had at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
Number analyzed (Participants) | 17 | 16 | 2 | 12 | 9
Participants
  PR interval value >=300 msec | 0 | 0 | 0 | 0 | 0
  PR interval %change >=25/50% msec | 0 | 0 | 0 | 0 | 0
  QRS interval value >= 140 msec | 0 | 0 | 0 | 0 | 0
  QRS interval %change >=50% msec | 0 | 0 | 0 | 0 | 0
  QTcF 450 msec < value <=480 msec | 0 | 0 | 0 | 1 | 0
  QTcF 480 msec < value <=500 msec | 0 | 0 | 0 | 0 | 0
  QTcF value >500 msec | 0 | 0 | 0 | 0 | 0
  QTcF 30 msec < change <=60 msec | 0 | 0 | 0 | 0 | 0
  QTcF change >60 msec | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: (Part A) Number of Participants With Categorical Scores on the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS was an interview-based rating scale to systematically assess suicidal ideation and suicidal behavior. C-SSRS assessed whether participant experienced any of the following 1: completed suicide, 2: suicide attempt (response of "yes" on "actual attempt"), 3: preparatory acts toward imminent suicidal behavior ("yes" on "aborted attempt", "interrupted attempt", "preparatory acts or behavior"), 4: any suicidal behavior or ideation, suicidal ideation ("yes" on "wish to be dead", "non-specific active suicidal thoughts"), 7: self-injurious behavior, no suicidal intent ("yes" on "has participant engaged in non-suicidal self-injurious behavior").
Time Frame: Study Day -1 (D-1) (ie, Period 1 Day-1 [P1D-1]), D5 (P3D1), D12 (P3D8), D19 (P3D15), D27 (P3D23), D36 (P4D1), D40 (P6D1), D48 (P6D9), D58 (P6D19), D62 (P8D1), and at follow-up visit (Days 69-72) of Part A.
Population: The analysis set included all participants assigned to study intervention and who took at least 1 dose of study intervention. Participants with evaluable C-SSRS results were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants in Part A
Number analyzed (Participants) | 18
Participants
  Period 1 Day -1 / Atorvastatin 20 mg | 0
  Period 1 Day -1 / Atorvastatin 20 mg Past 12 Months | 0
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID (Since Last Visit): number analyzed (Participants) | 17
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID (Since Last Visit) | 0
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID (Since Last Visit): number analyzed (Participants) | 16
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID (Since Last Visit) | 0
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID (Since Last Visit): number analyzed (Participants) | 16
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID (Since Last Visit) | 0
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID (Since Last Visit): number analyzed (Participants) | 15
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID (Since Last Visit) | 0
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg (Since Last Visit): number analyzed (Participants) | 13
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg (Since Last Visit) | 0
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID (Since Last Visit): number analyzed (Participants) | 13
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID (Since Last Visit) | 0
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID (Since Last Visit): number analyzed (Participants) | 13
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID (Since Last Visit) | 0
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID (Since Last Visit): number analyzed (Participants) | 6
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID (Since Last Visit) | 0
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg (Since Last Visit): number analyzed (Participants) | 6
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg (Since Last Visit) | 0
  Follow Up (Since Last Visit): number analyzed (Participants) | 15
  Follow Up (Since Last Visit) | 0

16. Secondary Outcome: (Part B) Number of Participants With Categorical Scores on the C-SSRS
Description: as for outcome 15
Time Frame: Study Day -1 (D-1) (ie, Period 1 Day-1 [P1D-1]), D6 (P2D1), D13 (P2D8), D20 (P2D15), D27 (P2D22), D37 (P3D1), D42 (P4D1), D50 (P4D9), D60 (P4D19), D66 (P5D6), and at follow-up visit (Days 72-75) of Part B.
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants in Part B
Number analyzed (Participants) | 17
Participants
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE | 0
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE (Past 12 months) | 0
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID (Since Last Visit): number analyzed (Participants) | 16
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID (Since Last Visit) | 0
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID (Since Last Visit): number analyzed (Participants) | 16
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID (Since Last Visit) | 0
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID (Since Last Visit): number analyzed (Participants) | 16
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID (Since Last Visit) | 0
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID (Since Last Visit): number analyzed (Participants) | 16
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID (Since Last Visit) | 0
  Period 3 Day 1 / PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Since Last Visit): number analyzed (Participants) | 15
  Period 3 Day 1 / PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Since Last Visit) | 0
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID (Since Last Visit): number analyzed (Participants) | 12
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID (Since Last Visit) | 0
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID (Since Last Visit): number analyzed (Participants) | 11
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID (Since Last Visit) | 0
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID (Since Last Visit): number analyzed (Participants) | 9
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID (Since Last Visit) | 0
  Period 5 Day 6 / PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Since Last Visit): number analyzed (Participants) | 9
  Period 5 Day 6 / PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Since Last Visit) | 0
  Follow Up (Since Last Visit): number analyzed (Participants) | 11
  Follow Up (Since Last Visit) | 0

17. Secondary Outcome: (Part A) Number of Participants With Categorical Scores on the Patient Health Questionnaire (PHQ-9)
Description: The PHQ-9 is a 9 item self-report scale for the assessment of depressive symptoms. The questions included "little interest/pleasure in things", "feeling down depressed or hopeless", "trouble falling or staying asleep", "feeling tired or little energy", "poor appetite or overeating", "feeling bad about yourself", "trouble concentrating on things", "moving slowly or fidgety/restless" and "thoughts you be better off dead". Each item was scored on scale of "not at all", "several days", "more than half the days" to "nearly every day". Total score range: 0-27 (each item with scale from 0 [not at all] to 3 [nearly every day]. Higher score=greater severity).
Time Frame: as for outcome 15
Population: The analysis set included all participants assigned to study intervention and who took at least 1 dose of study intervention. Participants with evaluable PHQ-9 results were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants in Part A
Number analyzed (Participants) | 18
Participants
  Period 1 Day -1 / Atorvastatin 20 mg / Little Interest/Pleasure in Things: Not At All | 18
  Period 1 Day -1 / Atorvastatin 20 mg / Little Interest/Pleasure in Things: Several Days | 0
  Period 1 Day -1 / Atorvastatin 20 mg / Little Interest/Pleasure in Things: More Than Half The Days | 0
  Period 1 Day -1 / Atorvastatin 20 mg / Little Interest/Pleasure in Things: Nearly Every Day | 0
  Period 1 Day -1 / Atorvastatin 20 mg / Feeling Down Depressed or Hopeless: Not At All | 18
  Period 1 Day -1 / Atorvastatin 20 mg / Feeling Down Depressed or Hopeless: Several Days | 0
  Period 1 Day -1 / Atorvastatin 20 mg / Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Period 1 Day -1 / Atorvastatin 20 mg / Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Period 1 Day -1 / Atorvastatin 20 mg / Trouble Falling or Staying Asleep: Not At All | 18
  Period 1 Day -1 / Atorvastatin 20 mg / Trouble Falling or Staying Asleep: Several Days | 0
  Period 1 Day -1 / Atorvastatin 20 mg / Trouble Falling or Staying Asleep: More Than Half The Days | 0
  Period 1 Day -1 / Atorvastatin 20 mg / Trouble Falling or Staying Asleep: Nearly Every Day | 0
  Period 1 Day -1 / Atorvastatin 20 mg / Feeling Tired or Little Energy: Not At All | 18
  Period 1 Day -1 / Atorvastatin 20 mg / Feeling Tired or Little Energy: Several Days | 0
  Period 1 Day -1 / Atorvastatin 20 mg / Feeling Tired or Little Energy: More Than Half The Days | 0
  Period 1 Day -1 / Atorvastatin 20 mg / Feeling Tired or Little Energy: Nearly Every Day | 0
  Period 1 Day -1 / Atorvastatin 20 mg / Poor Appetite or Overeating: Not At All | 18
  Period 1 Day -1 / Atorvastatin 20 mg / Poor Appetite or Overeating: Several Days | 0
  Period 1 Day -1 / Atorvastatin 20 mg / Poor Appetite or Overeating: More Than Half The Days | 0
  Period 1 Day -1 / Atorvastatin 20 mg / Poor Appetite or Overeating: Nearly Every Day | 0
  Period 1 Day -1 / Atorvastatin 20 mg / Feeling Bad About Yourself: Not At All | 18
  Period 1 Day -1 / Atorvastatin 20 mg / Feeling Bad About Yourself: Several Days | 0
  Period 1 Day -1 / Atorvastatin 20 mg / Feeling Bad About Yourself: More Than Half The Days | 0
  Period 1 Day -1 / Atorvastatin 20 mg / Feeling Bad About Yourself: Nearly Every Day | 0
  Period 1 Day -1 / Atorvastatin 20 mg / Trouble Concentrating on Things: Not At All | 18
  Period 1 Day -1 / Atorvastatin 20 mg / Trouble Concentrating on Things: Several Days | 0
  Period 1 Day -1 / Atorvastatin 20 mg / Trouble Concentrating on Things: More Than Half The Days | 0
  Period 1 Day -1 / Atorvastatin 20 mg / Trouble Concentrating on Things: Nearly Every Day | 0
  Period 1 Day -1 / Atorvastatin 20 mg / Moving Slowly or Fidgety/Restless: Not At All | 18
  Period 1 Day -1 / Atorvastatin 20 mg / Moving Slowly or Fidgety/Restless: Several Days | 0
  Period 1 Day -1 / Atorvastatin 20 mg / Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  Period 1 Day -1 / Atorvastatin 20 mg / Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  Period 1 Day -1 / Atorvastatin 20 mg / Thoughts You Be Better Off Dead: Not At All | 18
  Period 1 Day -1 / Atorvastatin 20 mg / Thoughts You Be Better Off Dead: Several Days | 0
  Period 1 Day -1 / Atorvastatin 20 mg / Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Period 1 Day -1 / Atorvastatin 20 mg / Thoughts You Be Better Off Dead: Nearly Every Day | 0
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: number analyzed (Participants) | 17
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: Not At All | 17
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: Several Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: More Than Half The Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: Nearly Every Day | 0
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: number analyzed (Participants) | 17
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: Not At All | 17
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: Several Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: number analyzed (Participants) | 17
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: Not At All | 17
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: Several Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: More Than Half The Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: Nearly Every Day | 0
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: number analyzed (Participants) | 17
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: Not At All | 17
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: Several Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: More Than Half The Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: Nearly Every Day | 0
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: number analyzed (Participants) | 17
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: Not At All | 17
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: Several Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: More Than Half The Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: Nearly Every Day | 0
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: number analyzed (Participants) | 17
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: Not At All | 17
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: Several Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: More Than Half The Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: Nearly Every Day | 0
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: number analyzed (Participants) | 17
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: Not At All | 17
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: Several Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: More Than Half The Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: Nearly Every Day | 0
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: number analyzed (Participants) | 17
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: Not At All | 17
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: Several Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: number analyzed (Participants) | 17
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: Not At All | 17
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: Several Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: Nearly Every Day | 0
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: number analyzed (Participants) | 16
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: Not At All | 16
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: Several Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: More Than Half The Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: Nearly Every Day | 0
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: number analyzed (Participants) | 16
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: Not At All | 16
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: Several Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: number analyzed (Participants) | 16
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: Not At All | 16
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: Several Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: More Than Half The Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: Nearly Every Day | 0
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: number analyzed (Participants) | 16
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: Not At All | 16
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: Several Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: More Than Half The Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: Nearly Every Day | 0
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: number analyzed (Participants) | 16
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: Not At All | 15
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: Several Days | 1
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: More Than Half The Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: Nearly Every Day | 0
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: number analyzed (Participants) | 16
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: Not At All | 16
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: Several Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: More Than Half The Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: Nearly Every Day | 0
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: number analyzed (Participants) | 16
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: Not At All | 16
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: Several Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: More Than Half The Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: Nearly Every Day | 0
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: number analyzed (Participants) | 16
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: Not At All | 16
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: Several Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: number analyzed (Participants) | 16
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: Not At All | 16
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: Several Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: Nearly Every Day | 0
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: number analyzed (Participants) | 16
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: Not At All | 16
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: Several Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: More Than Half The Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: Nearly Every Day | 0
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: number analyzed (Participants) | 16
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: Not At All | 16
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: Several Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: number analyzed (Participants) | 16
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: Not At All | 16
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: Several Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: More Than Half The Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: Nearly Every Day | 0
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: number analyzed (Participants) | 16
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: Not At All | 16
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: Several Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: More Than Half The Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: Nearly Every Day | 0
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: number analyzed (Participants) | 16
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: Not At All | 15
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: Several Days | 1
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: More Than Half The Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: Nearly Every Day | 0
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: number analyzed (Participants) | 16
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: Not At All | 16
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: Several Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: More Than Half The Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: Nearly Every Day | 0
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: number analyzed (Participants) | 16
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: Not At All | 16
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: Several Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: More Than Half The Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: Nearly Every Day | 0
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: number analyzed (Participants) | 16
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: Not At All | 16
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: Several Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: number analyzed (Participants) | 16
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: Not At All | 16
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: Several Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: Nearly Every Day | 0
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: number analyzed (Participants) | 15
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: Not At All | 15
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: Several Days | 0
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: More Than Half The Days | 0
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: Nearly Every Day | 0
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: number analyzed (Participants) | 15
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: Not At All | 15
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: Several Days | 0
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: number analyzed (Participants) | 15
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: Not At All | 15
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: Several Days | 0
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: More Than Half The Days | 0
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: Nearly Every Day | 0
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: number analyzed (Participants) | 15
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: Not At All | 15
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: Several Days | 0
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: More Than Half The Days | 0
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: Nearly Every Day | 0
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: number analyzed (Participants) | 15
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: Not At All | 12
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: Several Days | 1
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: More Than Half The Days | 1
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: Nearly Every Day | 1
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: number analyzed (Participants) | 15
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: Not At All | 15
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: Several Days | 0
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: More Than Half The Days | 0
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: Nearly Every Day | 0
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: number analyzed (Participants) | 15
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: Not At All | 15
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: Several Days | 0
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: More Than Half The Days | 0
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: Nearly Every Day | 0
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: number analyzed (Participants) | 15
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: Not At All | 15
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: Several Days | 0
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: number analyzed (Participants) | 15
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: Not At All | 15
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: Several Days | 0
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Period 3 Day 23 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: Nearly Every Day | 0
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Little Interest/Pleasure in Things: number analyzed (Participants) | 13
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Little Interest/Pleasure in Things: Not At All | 13
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Little Interest/Pleasure in Things: Several Days | 0
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Little Interest/Pleasure in Things: More Than Half The Days | 0
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Little Interest/Pleasure in Things: Nearly Every Day | 0
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Feeling Down Depressed or Hopeless: number analyzed (Participants) | 13
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Feeling Down Depressed or Hopeless: Not At All | 13
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Feeling Down Depressed or Hopeless: Several Days | 0
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Trouble Falling or Staying Asleep: number analyzed (Participants) | 13
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Trouble Falling or Staying Asleep: Not At All | 13
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Trouble Falling or Staying Asleep: Several Days | 0
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Trouble Falling or Staying Asleep: More Than Half The Days | 0
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Trouble Falling or Staying Asleep: Nearly Every Day | 0
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Feeling Tired or Little Energy: number analyzed (Participants) | 13
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Feeling Tired or Little Energy: Not At All | 13
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Feeling Tired or Little Energy: Several Days | 0
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Feeling Tired or Little Energy: More Than Half The Days | 0
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Feeling Tired or Little Energy: Nearly Every Day | 0
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Poor Appetite or Overeating: number analyzed (Participants) | 13
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Poor Appetite or Overeating: Not At All | 10
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Poor Appetite or Overeating: Several Days | 2
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Poor Appetite or Overeating: More Than Half The Days | 0
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Poor Appetite or Overeating: Nearly Every Day | 1
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Feeling Bad About Yourself: number analyzed (Participants) | 13
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Feeling Bad About Yourself: Not At All | 13
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Feeling Bad About Yourself: Several Days | 0
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Feeling Bad About Yourself: More Than Half The Days | 0
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Feeling Bad About Yourself: Nearly Every Day | 0
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Trouble Concentrating on Things: number analyzed (Participants) | 13
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Trouble Concentrating on Things: Not At All | 13
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Trouble Concentrating on Things: Several Days | 0
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Trouble Concentrating on Things: More Than Half The Days | 0
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Trouble Concentrating on Things: Nearly Every Day | 0
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Moving Slowly or Fidgety/Restless: number analyzed (Participants) | 13
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Moving Slowly or Fidgety/Restless: Not At All | 13
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Moving Slowly or Fidgety/Restless: Several Days | 0
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Thoughts You Be Better Off Dead: number analyzed (Participants) | 13
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Thoughts You Be Better Off Dead: Not At All | 13
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Thoughts You Be Better Off Dead: Several Days | 0
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Period 4 Day 1 / PF-06882961 120 mg BID + Atorvastatin 20 mg / Thoughts You Be Better Off Dead: Nearly Every Day | 0
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Little Interest/Pleasure in Things: number analyzed (Participants) | 13
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Little Interest/Pleasure in Things: Not At All | 13
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Little Interest/Pleasure in Things: Several Days | 0
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Little Interest/Pleasure in Things: More Than Half The Days | 0
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Little Interest/Pleasure in Things: Nearly Every Day | 0
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Feeling Down Depressed or Hopeless: number analyzed (Participants) | 13
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Feeling Down Depressed or Hopeless: Not At All | 13
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Feeling Down Depressed or Hopeless: Several Days | 0
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Trouble Falling or Staying Asleep: number analyzed (Participants) | 13
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Trouble Falling or Staying Asleep: Not At All | 12
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Trouble Falling or Staying Asleep: Several Days | 0
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Trouble Falling or Staying Asleep: More Than Half The Days | 1
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Trouble Falling or Staying Asleep: Nearly Every Day | 0
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Feeling Tired or Little Energy: number analyzed (Participants) | 13
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Feeling Tired or Little Energy: Not At All | 12
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Feeling Tired or Little Energy: Several Days | 1
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Feeling Tired or Little Energy: More Than Half The Days | 0
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Feeling Tired or Little Energy: Nearly Every Day | 0
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Poor Appetite or Overeating: number analyzed (Participants) | 13
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Poor Appetite or Overeating: Not At All | 8
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Poor Appetite or Overeating: Several Days | 2
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Poor Appetite or Overeating: More Than Half The Days | 1
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Poor Appetite or Overeating: Nearly Every Day | 2
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Feeling Bad About Yourself: number analyzed (Participants) | 13
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Feeling Bad About Yourself: Not At All | 13
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Feeling Bad About Yourself: Several Days | 0
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Feeling Bad About Yourself: More Than Half The Days | 0
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Feeling Bad About Yourself: Nearly Every Day | 0
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Trouble Concentrating on Things: number analyzed (Participants) | 13
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Trouble Concentrating on Things: Not At All | 13
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Trouble Concentrating on Things: Several Days | 0
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Trouble Concentrating on Things: More Than Half The Days | 0
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Trouble Concentrating on Things: Nearly Every Day | 0
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Moving Slowly or Fidgety/Restless: number analyzed (Participants) | 13
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Moving Slowly or Fidgety/Restless: Not At All | 13
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Moving Slowly or Fidgety/Restless: Several Days | 0
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Thoughts You Be Better Off Dead: number analyzed (Participants) | 13
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Thoughts You Be Better Off Dead: Not At All | 13
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Thoughts You Be Better Off Dead: Several Days | 0
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID / Thoughts You Be Better Off Dead: Nearly Every Day | 0
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Little Interest/Pleasure in Things: number analyzed (Participants) | 13
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Little Interest/Pleasure in Things: Not At All | 11
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Little Interest/Pleasure in Things: Several Days | 2
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Little Interest/Pleasure in Things: More Than Half The Days | 0
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Little Interest/Pleasure in Things: Nearly Every Day | 0
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Feeling Down Depressed or Hopeless: number analyzed (Participants) | 13
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Feeling Down Depressed or Hopeless: Not At All | 13
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Feeling Down Depressed or Hopeless: Several Days | 0
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Trouble Falling or Staying Asleep: number analyzed (Participants) | 13
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Trouble Falling or Staying Asleep: Not At All | 11
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Trouble Falling or Staying Asleep: Several Days | 1
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Trouble Falling or Staying Asleep: More Than Half The Days | 0
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Trouble Falling or Staying Asleep: Nearly Every Day | 1
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID /Feeling Tired or Little Energy: number analyzed (Participants) | 13
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID /Feeling Tired or Little Energy: Not At All | 10
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID /Feeling Tired or Little Energy: Several Days | 2
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID /Feeling Tired or Little Energy: More Than Half The Days | 1
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID /Feeling Tired or Little Energy: Nearly Every Day | 0
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Poor Appetite or Overeating: number analyzed (Participants) | 13
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Poor Appetite or Overeating: Not At All | 7
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Poor Appetite or Overeating: Several Days | 2
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Poor Appetite or Overeating: More Than Half The Days | 1
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Poor Appetite or Overeating: Nearly Every Day | 3
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Feeling Bad About Yourself: number analyzed (Participants) | 13
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Feeling Bad About Yourself: Not At All | 13
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Feeling Bad About Yourself: Several Days | 0
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Feeling Bad About Yourself: More Than Half The Days | 0
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Feeling Bad About Yourself: Nearly Every Day | 0
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Trouble Concentrating on Things: number analyzed (Participants) | 13
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Trouble Concentrating on Things: Not At All | 13
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Trouble Concentrating on Things: Several Days | 0
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Trouble Concentrating on Things: More Than Half The Days | 0
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Trouble Concentrating on Things: Nearly Every Day | 0
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Moving Slowly or Fidgety/Restless: number analyzed (Participants) | 13
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Moving Slowly or Fidgety/Restless: Not At All | 13
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Moving Slowly or Fidgety/Restless: Several Days | 0
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Thoughts You Be Better Off Dead: number analyzed (Participants) | 13
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Thoughts You Be Better Off Dead: Not At All | 13
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Thoughts You Be Better Off Dead: Several Days | 0
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID / Thoughts You Be Better Off Dead: Nearly Every Day | 0
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Little Interest/Pleasure in Things: number analyzed (Participants) | 6
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Little Interest/Pleasure in Things: Not At All | 5
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Little Interest/Pleasure in Things: Several Days | 1
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Little Interest/Pleasure in Things: More Than Half The Days | 0
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Little Interest/Pleasure in Things: Nearly Every Day | 0
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Feeling Down Depressed or Hopeless: number analyzed (Participants) | 6
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Feeling Down Depressed or Hopeless: Not At All | 6
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Feeling Down Depressed or Hopeless: Several Days | 0
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Trouble Falling or Staying Asleep: number analyzed (Participants) | 6
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Trouble Falling or Staying Asleep: Not At All | 5
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Trouble Falling or Staying Asleep: Several Days | 1
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Trouble Falling or Staying Asleep: More Than Half The Days | 0
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Trouble Falling or Staying Asleep: Nearly Every Day | 0
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Feeling Tired or Little Energy: number analyzed (Participants) | 6
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Feeling Tired or Little Energy: Not At All | 5
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Feeling Tired or Little Energy: Several Days | 0
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Feeling Tired or Little Energy: More Than Half The Days | 1
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Feeling Tired or Little Energy: Nearly Every Day | 0
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Poor Appetite or Overeating: number analyzed (Participants) | 6
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Poor Appetite or Overeating: Not At All | 5
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Poor Appetite or Overeating: Several Days | 0
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Poor Appetite or Overeating: More Than Half The Days | 1
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Poor Appetite or Overeating: Nearly Every Day | 0
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Feeling Bad About Yourself: number analyzed (Participants) | 6
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Feeling Bad About Yourself: Not At All | 6
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Feeling Bad About Yourself: Several Days | 0
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Feeling Bad About Yourself: More Than Half The Days | 0
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Feeling Bad About Yourself: Nearly Every Day | 0
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Trouble Concentrating on Things: number analyzed (Participants) | 6
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Trouble Concentrating on Things: Not At All | 5
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Trouble Concentrating on Things: Several Days | 1
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Trouble Concentrating on Things: More Than Half The Days | 0
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Trouble Concentrating on Things: Nearly Every Day | 0
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Moving Slowly or Fidgety/Restless: number analyzed (Participants) | 6
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Moving Slowly or Fidgety/Restless: Not At All | 5
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Moving Slowly or Fidgety/Restless: Several Days | 1
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Thoughts You Be Better Off Dead: number analyzed (Participants) | 6
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Thoughts You Be Better Off Dead: Not At All | 6
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Thoughts You Be Better Off Dead: Several Days | 0
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Period 6 Day 19 / PF-06882961 titration up to 200 mg BID / Thoughts You Be Better Off Dead: Nearly Every Day | 0
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Little Interest/Pleasure in Things: number analyzed (Participants) | 6
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Little Interest/Pleasure in Things: Not At All | 5
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Little Interest/Pleasure in Things: Several Days | 1
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Little Interest/Pleasure in Things: More Than Half The Days | 0
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Little Interest/Pleasure in Things: Nearly Every Day | 0
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Feeling Down Depressed or Hopeless: number analyzed (Participants) | 6
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Feeling Down Depressed or Hopeless: Not At All | 5
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Feeling Down Depressed or Hopeless: Several Days | 1
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Trouble Falling or Staying Asleep: number analyzed (Participants) | 6
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Trouble Falling or Staying Asleep: Not At All | 5
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Trouble Falling or Staying Asleep: Several Days | 1
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Trouble Falling or Staying Asleep: More Than Half The Days | 0
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Trouble Falling or Staying Asleep: Nearly Every Day | 0
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Feeling Tired or Little Energy: number analyzed (Participants) | 6
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Feeling Tired or Little Energy: Not At All | 5
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Feeling Tired or Little Energy: Several Days | 1
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Feeling Tired or Little Energy: More Than Half The Days | 0
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Feeling Tired or Little Energy: Nearly Every Day | 0
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Poor Appetite or Overeating: number analyzed (Participants) | 6
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Poor Appetite or Overeating: Not At All | 5
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Poor Appetite or Overeating: Several Days | 0
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Poor Appetite or Overeating: More Than Half The Days | 1
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Poor Appetite or Overeating: Nearly Every Day | 0
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Feeling Bad About Yourself: number analyzed (Participants) | 6
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Feeling Bad About Yourself: Not At All | 6
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Feeling Bad About Yourself: Several Days | 0
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Feeling Bad About Yourself: More Than Half The Days | 0
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Feeling Bad About Yourself: Nearly Every Day | 0
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Trouble Concentrating on Things: number analyzed (Participants) | 6
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Trouble Concentrating on Things: Not At All | 5
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Trouble Concentrating on Things: Several Days | 1
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Trouble Concentrating on Things: More Than Half The Days | 0
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Trouble Concentrating on Things: Nearly Every Day | 0
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Moving Slowly or Fidgety/Restless: number analyzed (Participants) | 6
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Moving Slowly or Fidgety/Restless: Not At All | 5
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Moving Slowly or Fidgety/Restless: Several Days | 1
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Thoughts You Be Better Off Dead: number analyzed (Participants) | 6
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Thoughts You Be Better Off Dead: Not At All | 6
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Thoughts You Be Better Off Dead: Several Days | 0
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Period 8 Day 1 / PF-06882961 200 mg BID + Midazolam 5 mg / Thoughts You Be Better Off Dead: Nearly Every Day | 0
  Follow Up: number analyzed (Participants) | 15
  Follow Up: Not At All | 14
  Follow Up: Several Days | 1
  Follow Up: More Than Half The Days | 0
  Follow Up: Nearly Every Day | 0

18. Secondary Outcome: (Part B) Number of Participants With Categorical Scores on the PHQ-9
Description: as for outcome 17
Time Frame: as for outcome 16
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants in Part B
Number analyzed (Participants) | 17
Participants
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Little Interest/Pleasure in Things: Not At All | 17
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Little Interest/Pleasure in Things: Several Days | 0
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Little Interest/Pleasure in Things: More Than Half The Days | 0
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Little Interest/Pleasure in Things: Nearly Every Day | 0
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Feeling Down Depressed or Hopeless: Not At All | 16
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Feeling Down Depressed or Hopeless: Several Days | 1
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Trouble Falling or Staying Asleep: Not At All | 17
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Trouble Falling or Staying Asleep: Several Days | 0
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Trouble Falling or Staying Asleep: More Than Half The Days | 0
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Trouble Falling or Staying Asleep: Nearly Every Day | 0
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Feeling Tired or Little Energy: Not At All | 16
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Feeling Tired or Little Energy: Several Days | 1
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Feeling Tired or Little Energy: More Than Half The Days | 0
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Feeling Tired or Little Energy: Nearly Every Day | 0
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Poor Appetite or Overeating: Not At All | 16
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Poor Appetite or Overeating: Several Days | 1
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Poor Appetite or Overeating: More Than Half The Days | 0
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Poor Appetite or Overeating: Nearly Every Day | 0
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Feeling Bad About Yourself: Not At All | 16
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Feeling Bad About Yourself: Several Days | 1
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Feeling Bad About Yourself: More Than Half The Days | 0
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Feeling Bad About Yourself: Nearly Every Day | 0
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Trouble Concentrating on Things: Not At All | 17
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Trouble Concentrating on Things: Several Days | 0
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Trouble Concentrating on Things: More Than Half The Days | 0
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Trouble Concentrating on Things: Nearly Every Day | 0
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Moving Slowly or Fidgety/Restless: Not At All | 17
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Moving Slowly or Fidgety/Restless: Several Days | 0
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Thoughts You Be Better Off Dead: Not At All | 17
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Thoughts You Be Better Off Dead: Several Days | 0
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Period 1 Day -1 / 0.15 mg LE & 0.03 mg EE / Thoughts You Be Better Off Dead: Nearly Every Day | 0
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: number analyzed (Participants) | 16
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: Not At All | 16
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: Several Days | 0
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: More Than Half The Days | 0
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: Nearly Every Day | 0
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: number analyzed (Participants) | 16
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: Not At All | 16
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: Several Days | 0
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: number analyzed (Participants) | 16
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: Not At All | 16
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: Several Days | 0
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: More Than Half The Days | 0
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: Nearly Every Day | 0
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: number analyzed (Participants) | 16
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: Not At All | 15
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: Several Days | 1
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: More Than Half The Days | 0
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: Nearly Every Day | 0
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: number analyzed (Participants) | 16
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: Not At All | 15
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: Several Days | 1
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: More Than Half The Days | 0
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: Nearly Every Day | 0
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: number analyzed (Participants) | 16
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: Not At All | 15
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: Several Days | 1
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: More Than Half The Days | 0
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: Nearly Every Day | 0
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: number analyzed (Participants) | 16
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: Not At All | 15
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: Several Days | 1
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: More Than Half The Days | 0
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: Nearly Every Day | 0
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: number analyzed (Participants) | 16
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: Not At All | 16
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: Several Days | 0
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: number analyzed (Participants) | 16
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: Not At All | 16
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: Several Days | 0
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Period 2 Day 1 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: Nearly Every Day | 0
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: number analyzed (Participants) | 16
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: Not At All | 16
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: Several Days | 0
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: More Than Half The Days | 0
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: Nearly Every Day | 0
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: number analyzed (Participants) | 16
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: Not At All | 16
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: Several Days | 0
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: number analyzed (Participants) | 16
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: Not At All | 16
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: Several Days | 0
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: More Than Half The Days | 0
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: Nearly Every Day | 0
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: number analyzed (Participants) | 16
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: Not At All | 15
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: Several Days | 1
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: More Than Half The Days | 0
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: Nearly Every Day | 0
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: number analyzed (Participants) | 16
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: Not At All | 15
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: Several Days | 1
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: More Than Half The Days | 0
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: Nearly Every Day | 0
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: number analyzed (Participants) | 16
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: Not At All | 16
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: Several Days | 0
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: More Than Half The Days | 0
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: Nearly Every Day | 0
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: number analyzed (Participants) | 16
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: Not At All | 16
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: Several Days | 0
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: More Than Half The Days | 0
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: Nearly Every Day | 0
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: number analyzed (Participants) | 16
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: Not At All | 16
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: Several Days | 0
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: number analyzed (Participants) | 16
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: Not At All | 16
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: Several Days | 0
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Period 2 Day 8 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: Nearly Every Day | 0
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: number analyzed (Participants) | 16
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: Not At All | 15
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: Several Days | 1
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: More Than Half The Days | 0
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: Nearly Every Day | 0
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: number analyzed (Participants) | 16
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: Not At All | 16
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: Several Days | 0
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: number analyzed (Participants) | 16
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: Not At All | 16
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: Several Days | 0
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: More Than Half The Days | 0
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: Nearly Every Day | 0
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: number analyzed (Participants) | 16
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: Not At All | 15
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: Several Days | 1
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: More Than Half The Days | 0
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: Nearly Every Day | 0
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: number analyzed (Participants) | 16
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: Not At All | 13
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: Several Days | 1
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: More Than Half The Days | 2
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: Nearly Every Day | 0
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: number analyzed (Participants) | 16
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: Not At All | 16
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: Several Days | 0
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: More Than Half The Days | 0
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: Nearly Every Day | 0
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: number analyzed (Participants) | 16
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: Not At All | 16
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: Several Days | 0
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: More Than Half The Days | 0
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: Nearly Every Day | 0
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: number analyzed (Participants) | 16
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: Not At All | 16
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: Several Days | 0
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: number analyzed (Participants) | 16
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: Not At All | 16
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: Several Days | 0
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Period 2 Day 15 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: Nearly Every Day | 0
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: number analyzed (Participants) | 16
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: Not At All | 15
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: Several Days | 1
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: More Than Half The Days | 0
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Little Interest/Pleasure in Things: Nearly Every Day | 0
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: number analyzed (Participants) | 16
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: Not At All | 16
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: Several Days | 0
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: number analyzed (Participants) | 16
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: Not At All | 16
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: Several Days | 0
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: More Than Half The Days | 0
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Trouble Falling or Staying Asleep: Nearly Every Day | 0
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: number analyzed (Participants) | 16
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: Not At All | 15
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: Several Days | 1
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: More Than Half The Days | 0
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Feeling Tired or Little Energy: Nearly Every Day | 0
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: number analyzed (Participants) | 16
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: Not At All | 13
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: Several Days | 3
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: More Than Half The Days | 0
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Poor Appetite or Overeating: Nearly Every Day | 0
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: number analyzed (Participants) | 16
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: Not At All | 16
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: Several Days | 0
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: More Than Half The Days | 0
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Feeling Bad About Yourself: Nearly Every Day | 0
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: number analyzed (Participants) | 16
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: Not At All | 16
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: Several Days | 0
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: More Than Half The Days | 0
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Trouble Concentrating on Things: Nearly Every Day | 0
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: number analyzed (Participants) | 16
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: Not At All | 16
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: Several Days | 0
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: number analyzed (Participants) | 16
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: Not At All | 16
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: Several Days | 0
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Period 2 Day 22 / PF-06882961 titration up to 120 mg BID / Thoughts You Be Better Off Dead: Nearly Every Day | 0
  Period 3 Day 1 / PF-06882961 120mg BID + 0.15mg LE & 0.03mg EE/Little Interest/Pleasure in Things: number analyzed (Participants) | 15
  Period 3 Day 1 / PF-06882961 120mg BID + 0.15mg LE & 0.03mg EE/Little Interest/Pleasure in Things: Not At All | 13
  Period 3 Day 1 / PF-06882961 120mg BID + 0.15mg LE & 0.03mg EE/Little Interest/Pleasure in Things: Several Days | 1
  Period 3 Day 1 / PF-06882961 120mg BID + 0.15mg LE & 0.03mg EE/Little Interest/Pleasure in Things: More Than Half The Days | 0
  Period 3 Day 1 / PF-06882961 120mg BID + 0.15mg LE & 0.03mg EE/Little Interest/Pleasure in Things: Nearly Every Day | 1
  Period 3 Day 1/PF-06882961 120mg BID + 0.15mg LE & 0.03mg EE/Feeling Down Depressed or Hopeless: number analyzed (Participants) | 15
  Period 3 Day 1/PF-06882961 120mg BID + 0.15mg LE & 0.03mg EE/Feeling Down Depressed or Hopeless: Not At All | 15
  Period 3 Day 1/PF-06882961 120mg BID + 0.15mg LE & 0.03mg EE/Feeling Down Depressed or Hopeless: Several Days | 0
  Period 3 Day 1/PF-06882961 120mg BID + 0.15mg LE & 0.03mg EE/Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Period 3 Day 1/PF-06882961 120mg BID + 0.15mg LE & 0.03mg EE/Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Period 3 Day 1/PF-06882961 120mg BID + 0.15mg LE & 0.03mg EE/Trouble Falling or Staying Asleep: number analyzed (Participants) | 15
  Period 3 Day 1/PF-06882961 120mg BID + 0.15mg LE & 0.03mg EE/Trouble Falling or Staying Asleep: Not At All | 14
  Period 3 Day 1/PF-06882961 120mg BID + 0.15mg LE & 0.03mg EE/Trouble Falling or Staying Asleep: Several Days | 0
  Period 3 Day 1/PF-06882961 120mg BID + 0.15mg LE & 0.03mg EE/Trouble Falling or Staying Asleep: More Than Half The Days | 1
  Period 3 Day 1/PF-06882961 120mg BID + 0.15mg LE & 0.03mg EE/Trouble Falling or Staying Asleep: Nearly Every Day | 0
  Period 3 Day 1 / PF-06882961 120mg BID + 0.15mg LE & 0.03mg EE/Feeling Tired or Little Energy: number analyzed (Participants) | 15
  Period 3 Day 1 / PF-06882961 120mg BID + 0.15mg LE & 0.03mg EE/Feeling Tired or Little Energy: Not At All | 13
  Period 3 Day 1 / PF-06882961 120mg BID + 0.15mg LE & 0.03mg EE/Feeling Tired or Little Energy: Several Days | 1
  Period 3 Day 1 / PF-06882961 120mg BID + 0.15mg LE & 0.03mg EE/Feeling Tired or Little Energy: More Than Half The Days | 0
  Period 3 Day 1 / PF-06882961 120mg BID + 0.15mg LE & 0.03mg EE/Feeling Tired or Little Energy: Nearly Every Day | 1
  Period 3 Day 1 / PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE / Poor Appetite or Overeating: number analyzed (Participants) | 15
  Period 3 Day 1 / PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE / Poor Appetite or Overeating: Not At All | 10
  Period 3 Day 1 / PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE / Poor Appetite or Overeating: Several Days | 0
  Period 3 Day 1 / PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE / Poor Appetite or Overeating: More Than Half The Days | 3
  Period 3 Day 1 / PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE / Poor Appetite or Overeating: Nearly Every Day | 2
  Period 3 Day 1 / PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE / Feeling Bad About Yourself: number analyzed (Participants) | 15
  Period 3 Day 1 / PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE / Feeling Bad About Yourself: Not At All | 15
  Period 3 Day 1 / PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE / Feeling Bad About Yourself: Several Days | 0
  Period 3 Day 1 / PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE / Feeling Bad About Yourself: More Than Half The Days | 0
  Period 3 Day 1 / PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE / Feeling Bad About Yourself: Nearly Every Day | 0
  Period 3 Day 1/PF-06882961 120mg BID + 0.15mg LE & 0.03mg EE/ Trouble Concentrating on Things: number analyzed (Participants) | 15
  Period 3 Day 1/PF-06882961 120mg BID + 0.15mg LE & 0.03mg EE/ Trouble Concentrating on Things: Not At All | 14
  Period 3 Day 1/PF-06882961 120mg BID + 0.15mg LE & 0.03mg EE/ Trouble Concentrating on Things: Several Days | 1
  Period 3 Day 1/PF-06882961 120mg BID + 0.15mg LE & 0.03mg EE/ Trouble Concentrating on Things: More Than Half The Days | 0
  Period 3 Day 1/PF-06882961 120mg BID + 0.15mg LE & 0.03mg EE/ Trouble Concentrating on Things: Nearly Every Day | 0
  Period 3 Day 1/PF-06882961 120mg BID + 0.15mg LE & 0.03mg EE/Moving Slowly or Fidgety/Restless: number analyzed (Participants) | 15
  Period 3 Day 1/PF-06882961 120mg BID + 0.15mg LE & 0.03mg EE/Moving Slowly or Fidgety/Restless: Not At All | 14
  Period 3 Day 1/PF-06882961 120mg BID + 0.15mg LE & 0.03mg EE/Moving Slowly or Fidgety/Restless: Several Days | 0
  Period 3 Day 1/PF-06882961 120mg BID + 0.15mg LE & 0.03mg EE/Moving Slowly or Fidgety/Restless: More Than Half The Days | 1
  Period 3 Day 1/PF-06882961 120mg BID + 0.15mg LE & 0.03mg EE/Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  Period 3 Day 1 / PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE / Thoughts You Be Better Off Dead: number analyzed (Participants) | 15
  Period 3 Day 1 / PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE / Thoughts You Be Better Off Dead: Not At All | 15
  Period 3 Day 1 / PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE / Thoughts You Be Better Off Dead: Several Days | 0
  Period 3 Day 1 / PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE / Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Period 3 Day 1 / PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE / Thoughts You Be Better Off Dead: Nearly Every Day | 0
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Little Interest/Pleasure in Things: number analyzed (Participants) | 12
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Little Interest/Pleasure in Things: Not At All | 11
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Little Interest/Pleasure in Things: Several Days | 1
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Little Interest/Pleasure in Things: More Than Half The Days | 0
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Little Interest/Pleasure in Things: Nearly Every Day | 0
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Feeling Down Depressed or Hopeless: number analyzed (Participants) | 12
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Feeling Down Depressed or Hopeless: Not At All | 12
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Feeling Down Depressed or Hopeless: Several Days | 0
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Trouble Falling or Staying Asleep: number analyzed (Participants) | 12
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Trouble Falling or Staying Asleep: Not At All | 12
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Trouble Falling or Staying Asleep: Several Days | 0
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Trouble Falling or Staying Asleep: More Than Half The Days | 0
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Trouble Falling or Staying Asleep: Nearly Every Day | 0
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Feeling Tired or Little Energy: number analyzed (Participants) | 12
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Feeling Tired or Little Energy: Not At All | 10
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Feeling Tired or Little Energy: Several Days | 2
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Feeling Tired or Little Energy: More Than Half The Days | 0
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Feeling Tired or Little Energy: Nearly Every Day | 0
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Poor Appetite or Overeating: number analyzed (Participants) | 12
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Poor Appetite or Overeating: Not At All | 9
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Poor Appetite or Overeating: Several Days | 0
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Poor Appetite or Overeating: More Than Half The Days | 1
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Poor Appetite or Overeating: Nearly Every Day | 2
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Feeling Bad About Yourself: number analyzed (Participants) | 12
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Feeling Bad About Yourself: Not At All | 12
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Feeling Bad About Yourself: Several Days | 0
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Feeling Bad About Yourself: More Than Half The Days | 0
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Feeling Bad About Yourself: Nearly Every Day | 0
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Trouble Concentrating on Things: number analyzed (Participants) | 12
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Trouble Concentrating on Things: Not At All | 12
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Trouble Concentrating on Things: Several Days | 0
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Trouble Concentrating on Things: More Than Half The Days | 0
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Trouble Concentrating on Things: Nearly Every Day | 0
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Moving Slowly or Fidgety/Restless: number analyzed (Participants) | 12
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Moving Slowly or Fidgety/Restless: Not At All | 12
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Moving Slowly or Fidgety/Restless: Several Days | 0
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Thoughts You Be Better Off Dead: number analyzed (Participants) | 12
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Thoughts You Be Better Off Dead: Not At All | 12
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Thoughts You Be Better Off Dead: Several Days | 0
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Period 4 Day 1 / PF-06882961 titration up to 200 mg BID / Thoughts You Be Better Off Dead: Nearly Every Day | 0
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Little Interest/Pleasure in Things: number analyzed (Participants) | 11
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Little Interest/Pleasure in Things: Not At All | 11
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Little Interest/Pleasure in Things: Several Days | 0
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Little Interest/Pleasure in Things: More Than Half The Days | 0
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Little Interest/Pleasure in Things: Nearly Every Day | 0
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Feeling Down Depressed or Hopeless: number analyzed (Participants) | 11
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Feeling Down Depressed or Hopeless: Not At All | 11
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Feeling Down Depressed or Hopeless: Several Days | 0
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Trouble Falling or Staying Asleep: number analyzed (Participants) | 11
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Trouble Falling or Staying Asleep: Not At All | 10
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Trouble Falling or Staying Asleep: Several Days | 1
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Trouble Falling or Staying Asleep: More Than Half The Days | 0
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Trouble Falling or Staying Asleep: Nearly Every Day | 0
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Feeling Tired or Little Energy: number analyzed (Participants) | 11
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Feeling Tired or Little Energy: Not At All | 10
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Feeling Tired or Little Energy: Several Days | 1
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Feeling Tired or Little Energy: More Than Half The Days | 0
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Feeling Tired or Little Energy: Nearly Every Day | 0
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Poor Appetite or Overeating: number analyzed (Participants) | 11
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Poor Appetite or Overeating: Not At All | 8
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Poor Appetite or Overeating: Several Days | 1
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Poor Appetite or Overeating: More Than Half The Days | 1
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Poor Appetite or Overeating: Nearly Every Day | 1
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Feeling Bad About Yourself: number analyzed (Participants) | 11
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Feeling Bad About Yourself: Not At All | 11
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Feeling Bad About Yourself: Several Days | 0
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Feeling Bad About Yourself: More Than Half The Days | 0
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Feeling Bad About Yourself: Nearly Every Day | 0
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Trouble Concentrating on Things: number analyzed (Participants) | 11
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Trouble Concentrating on Things: Not At All | 10
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Trouble Concentrating on Things: Several Days | 1
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Trouble Concentrating on Things: More Than Half The Days | 0
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Trouble Concentrating on Things: Nearly Every Day | 0
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Moving Slowly or Fidgety/Restless: number analyzed (Participants) | 11
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Moving Slowly or Fidgety/Restless: Not At All | 10
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Moving Slowly or Fidgety/Restless: Several Days | 1
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Thoughts You Be Better Off Dead: number analyzed (Participants) | 11
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Thoughts You Be Better Off Dead: Not At All | 11
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Thoughts You Be Better Off Dead: Several Days | 0
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Period 4 Day 9 / PF-06882961 titration up to 200 mg BID / Thoughts You Be Better Off Dead: Nearly Every Day | 0
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Little Interest/Pleasure in Things: number analyzed (Participants) | 9
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Little Interest/Pleasure in Things: Not At All | 9
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Little Interest/Pleasure in Things: Several Days | 0
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Little Interest/Pleasure in Things: More Than Half The Days | 0
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Little Interest/Pleasure in Things: Nearly Every Day | 0
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Feeling Down Depressed or Hopeless: number analyzed (Participants) | 9
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Feeling Down Depressed or Hopeless: Not At All | 9
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Feeling Down Depressed or Hopeless: Several Days | 0
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Trouble Falling or Staying Asleep: number analyzed (Participants) | 9
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Trouble Falling or Staying Asleep: Not At All | 8
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Trouble Falling or Staying Asleep: Several Days | 1
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Trouble Falling or Staying Asleep: More Than Half The Days | 0
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Trouble Falling or Staying Asleep: Nearly Every Day | 0
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Feeling Tired or Little Energy: number analyzed (Participants) | 9
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Feeling Tired or Little Energy: Not At All | 8
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Feeling Tired or Little Energy: Several Days | 0
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Feeling Tired or Little Energy: More Than Half The Days | 0
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Feeling Tired or Little Energy: Nearly Every Day | 1
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Poor Appetite or Overeating: number analyzed (Participants) | 9
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Poor Appetite or Overeating: Not At All | 7
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Poor Appetite or Overeating: Several Days | 0
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Poor Appetite or Overeating: More Than Half The Days | 1
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Poor Appetite or Overeating: Nearly Every Day | 1
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Feeling Bad About Yourself: number analyzed (Participants) | 9
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Feeling Bad About Yourself: Not At All | 9
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Feeling Bad About Yourself: Several Days | 0
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Feeling Bad About Yourself: More Than Half The Days | 0
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Feeling Bad About Yourself: Nearly Every Day | 0
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Trouble Concentrating on Things: number analyzed (Participants) | 9
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Trouble Concentrating on Things: Not At All | 8
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Trouble Concentrating on Things: Several Days | 0
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Trouble Concentrating on Things: More Than Half The Days | 1
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Trouble Concentrating on Things: Nearly Every Day | 0
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Moving Slowly or Fidgety/Restless: number analyzed (Participants) | 9
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Moving Slowly or Fidgety/Restless: Not At All | 8
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Moving Slowly or Fidgety/Restless: Several Days | 0
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Moving Slowly or Fidgety/Restless: Nearly Every Day | 1
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Thoughts You Be Better Off Dead: number analyzed (Participants) | 9
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Thoughts You Be Better Off Dead: Not At All | 9
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Thoughts You Be Better Off Dead: Several Days | 0
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Period 4 Day 19 / PF-06882961 titration up to 200 mg BID /Thoughts You Be Better Off Dead: Nearly Every Day | 0
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Little Interest/Pleasure in Things: number analyzed (Participants) | 9
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Little Interest/Pleasure in Things: Not At All | 9
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Little Interest/Pleasure in Things: Several Days | 0
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Little Interest/Pleasure in Things: More Than Half The Days | 0
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Little Interest/Pleasure in Things: Nearly Every Day | 0
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Feeling Down Depressed or Hopeless: number analyzed (Participants) | 9
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Feeling Down Depressed or Hopeless: Not At All | 9
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Feeling Down Depressed or Hopeless: Several Days | 0
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Trouble Falling or Staying Asleep: number analyzed (Participants) | 9
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Trouble Falling or Staying Asleep: Not At All | 8
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Trouble Falling or Staying Asleep: Several Days | 0
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Trouble Falling or Staying Asleep: More Than Half The Days | 0
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Trouble Falling or Staying Asleep: Nearly Every Day | 1
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Feeling Tired or Little Energy: number analyzed (Participants) | 9
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Feeling Tired or Little Energy: Not At All | 8
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Feeling Tired or Little Energy: Several Days | 0
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Feeling Tired or Little Energy: More Than Half The Days | 0
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Feeling Tired or Little Energy: Nearly Every Day | 1
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Poor Appetite or Overeating: number analyzed (Participants) | 9
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Poor Appetite or Overeating: Not At All | 7
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Poor Appetite or Overeating: Several Days | 0
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Poor Appetite or Overeating: More Than Half The Days | 1
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Poor Appetite or Overeating: Nearly Every Day | 1
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Feeling Bad About Yourself: number analyzed (Participants) | 9
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Feeling Bad About Yourself: Not At All | 9
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Feeling Bad About Yourself: Several Days | 0
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Feeling Bad About Yourself: More Than Half The Days | 0
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Feeling Bad About Yourself: Nearly Every Day | 0
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Trouble Concentrating on Things: number analyzed (Participants) | 9
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Trouble Concentrating on Things: Not At All | 8
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Trouble Concentrating on Things: Several Days | 0
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Trouble Concentrating on Things: More Than Half The Days | 0
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Trouble Concentrating on Things: Nearly Every Day | 1
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Moving Slowly or Fidgety/Restless: number analyzed (Participants) | 9
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Moving Slowly or Fidgety/Restless: Not At All | 8
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Moving Slowly or Fidgety/Restless: Several Days | 0
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  Period 5 Day 6/PF-06882961 200mg BID+0.15mg LE & 0.03mg EE/Moving Slowly or Fidgety/Restless: Nearly Every Day | 1
  Period 5 Day 6 / PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE / Thoughts You Be Better Off Dead: number analyzed (Participants) | 9
  Period 5 Day 6 / PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE / Thoughts You Be Better Off Dead: Not At All | 9
  Period 5 Day 6 / PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE / Thoughts You Be Better Off Dead: Several Days | 0
  Period 5 Day 6 / PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE / Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Period 5 Day 6 / PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE / Thoughts You Be Better Off Dead: Nearly Every Day | 0
  Follow Up / Little Interest/Pleasure in Things: number analyzed (Participants) | 11
  Follow Up / Little Interest/Pleasure in Things: Not At All | 11
  Follow Up / Little Interest/Pleasure in Things: Several Days | 0
  Follow Up / Little Interest/Pleasure in Things: More Than Half The Days | 0
  Follow Up / Little Interest/Pleasure in Things: Nearly Every Day | 0
  Follow Up / Feeling Down Depressed or Hopeless: number analyzed (Participants) | 11
  Follow Up / Feeling Down Depressed or Hopeless: Not At All | 11
  Follow Up / Feeling Down Depressed or Hopeless: Several Days | 0
  Follow Up / Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Follow Up / Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Follow Up / Trouble Falling or Staying Asleep: number analyzed (Participants) | 11
  Follow Up / Trouble Falling or Staying Asleep: Not At All | 10
  Follow Up / Trouble Falling or Staying Asleep: Several Days | 1
  Follow Up / Trouble Falling or Staying Asleep: More Than Half The Days | 0
  Follow Up / Trouble Falling or Staying Asleep: Nearly Every Day | 0
  Follow Up / Feeling Tired or Little Energy: number analyzed (Participants) | 11
  Follow Up / Feeling Tired or Little Energy: Not At All | 11
  Follow Up / Feeling Tired or Little Energy: Several Days | 0
  Follow Up / Feeling Tired or Little Energy: More Than Half The Days | 0
  Follow Up / Feeling Tired or Little Energy: Nearly Every Day | 0
  Follow Up / Poor Appetite or Overeating: number analyzed (Participants) | 11
  Follow Up / Poor Appetite or Overeating: Not At All | 11
  Follow Up / Poor Appetite or Overeating: Several Days | 0
  Follow Up / Poor Appetite or Overeating: More Than Half The Days | 0
  Follow Up / Poor Appetite or Overeating: Nearly Every Day | 0
  Follow Up / Feeling Bad About Yourself: number analyzed (Participants) | 11
  Follow Up / Feeling Bad About Yourself: Not At All | 11
  Follow Up / Feeling Bad About Yourself: Several Days | 0
  Follow Up / Feeling Bad About Yourself: More Than Half The Days | 0
  Follow Up / Feeling Bad About Yourself: Nearly Every Day | 0
  Follow Up / Trouble Concentrating on Things: number analyzed (Participants) | 11
  Follow Up / Trouble Concentrating on Things: Not At All | 11
  Follow Up / Trouble Concentrating on Things: Several Days | 0
  Follow Up / Trouble Concentrating on Things: More Than Half The Days | 0
  Follow Up / Trouble Concentrating on Things: Nearly Every Day | 0
  Follow Up / Moving Slowly or Fidgety/Restless: number analyzed (Participants) | 11
  Follow Up / Moving Slowly or Fidgety/Restless: Not At All | 11
  Follow Up / Moving Slowly or Fidgety/Restless: Several Days | 0
  Follow Up / Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  Follow Up / Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  Follow Up / Thoughts You Be Better Off Dead: number analyzed (Participants) | 11
  Follow Up / Thoughts You Be Better Off Dead: Not At All | 11
  Follow Up / Thoughts You Be Better Off Dead: Several Days | 0
  Follow Up / Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Follow Up / Thoughts You Be Better Off Dead: Nearly Every Day | 0

ADVERSE EVENTS:
Time Frame: From Screening (Days 28 to -2) to follow-up telephone contact (Days 90 to 97) in Part A and from Screening (Days 28 to -2) to follow-up telephone contact (Days 94 to 101) in Part B of the study.
Arm/Group | Atorvastatin 20 mg (Part A Period 1) | Midazolam 5 mg (Part A Period 2) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8) | 0.15 mg LE & 0.03 mg EE (Part B Period 1) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/17 | 0/13 | 0/13 | 0/13 | 0/5 | 0/6 | 0/17 | 0/16 | 0/14 | 0/12 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/17 | 0/13 | 0/13 | 0/13 | 0/5 | 0/6 | 0/17 | 0/16 | 0/14 | 0/12 | 0/9
Other Adverse Events (participants affected / at risk) | 2/18 | 3/18 | 13/17 | 5/13 | 4/13 | 12/13 | 5/5 | 2/6 | 5/17 | 15/16 | 7/14 | 12/12 | 7/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atorvastatin 20 mg (Part A Period 1) (N=18) | Midazolam 5 mg (Part A Period 2) (N=18) | PF-06882961 Titration up to 120 mg BID (Part A Period 3) (N=17) | PF-06882961 120 mg BID + Atorvastatin 20 mg (Part A Period 4) (N=13) | PF-06882961 120 mg BID + Midazolam 5 mg (Part A Period 5) (N=13) | PF-06882961 Titration up to 200 mg BID (Part A Period 6) (N=13) | PF-06882961 200 mg BID + Atorvastatin 20 mg (Part A Period 7) (N=5) | PF-06882961 200 mg BID + Midazolam 5 mg (Part A Period 8) (N=6) | 0.15 mg LE & 0.03 mg EE (Part B Period 1) (N=17) | PF-06882961 Titration up to 120 mg BID (Part B Period 2) (N=16) | PF-06882961 120 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 3) (N=14) | PF-06882961 Titration up to 200 mg BID (Part B Period 4) (N=12) | PF-06882961 200 mg BID + 0.15 mg LE & 0.03 mg EE (Part B Period 5) (N=9)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 5 | 0 | 1 | 2 | 0 | 0 | 0 | 7 | 1 | 4 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 6 | 3 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 10 | 2 | 1 | 3 | 0 | 0 | 0 | 12 | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 1 | 5 | 1 | 0 | 0 | 5 | 1 | 3 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 3 | 1 | 0 | 2 | 0 | 0 | 0 | 4 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 1 | 3 | 0
Headache (Nervous system disorders) | 1 | 1 | 3 | 0 | 0 | 3 | 1 | 1 | 1 | 7 | 3 | 6 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling jittery (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood calcitonin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 2 | 0 | 0 | 8 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Initial insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Middle insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Electric shock sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0
Self esteem decreased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
In part A, a majority of participants discontinued from study interventions due to SARS-CoV-2 infection and data from only 3 to 4 participants were evaluable following administration of danuglipron 200 mg BID. The resulting data should, therefore, be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/05/NCT05093205/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/05/NCT05093205/SAP_001.pdf